CLINICAL TRIAL: NCT06974994
Title: Resilience to Antibiotic-induced Obesogenic Microbiota Vertically Transferred to the Neonatal Gut: Discovering Mechanism of Microbiota Modulation
Brief Title: Resilience to Antibiotic-induced Obesogenic Microbiota: Discovering Mechanism of Microbiota Modulation
Acronym: ReCoverHealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Principal Investigator, Erika Isolauri, Professor of Paediatrics, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: T1927_2023
Record Dates: First submitted 2025-04-27; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy Newborn Infants
Keywords: antibiotics; human milk oligosaccharides; probiotics; newborn; microbiome; microbiota; obesity; infectious diseases
MeSH Terms: conditions — Obesity; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic (Active Comparator): Bifidobacterium bifidum and human milk oligosaccharides (HMOs)
  Interventions: Dietary Supplement: Synbiotic Supplement
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic Supplement — Bifidobacterium bifidum and human milk oligosaccharides (HMOs)
  Arms: Synbiotic
Other: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The aim is to study whether the microbiota of children who are exposed to antibiotics at birth could be modified by synbiotic supplement and thereby reduce the risk of obesity, chronic diseases and respiratory tract infections. A total of 125 mother-child pairs will be recruited in this randomized, double-blind, placebo-controlled study. Infants are randomized to receive either a synbiotic supplement or a placebo for 2 months, after which their growth and morbidity will be monitored at the research clinic for 2 years.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women (n=125) and their newborn children who receive antibiotic treatment at delivery.

Exclusion Criteria:

* Chorioamnionitis
* Pre-eclampsia and hepatogestosis
* Suspected malformation or serious condition of the foetus and neonates
* Serious infection or other conditions not permitting breast milk feeding

Min Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
BMI at 24 months of age | From enrollment to 24 months of age
  Child's body mass index (BMI) at the age of 24 months

SECONDARY OUTCOMES:
Height | From enrollment to 24 months of age
  Child's height at the age of 6, 12, 18, and 24 months
Weight | From enrollment to 24 months of age
  Child's weight at the age of 6, 12, 18, and 24 months
Growth velocity | From enrollment to 3 months of age
  Child's growth velocity at 2-3 months of age
Child's microbiome | From enrollment to 24 months of age
  The function and composition of the child's gut, nasal, and mouth microbiome at the age of 2, 6, 12, 18, and 24 months
Mother's microbiome | From enrollment to 6 months after giving birth
  The function and composition of the mother's gut, nasal, and mouth microbiome when the child is 2 and 6 months of age
Breast milk microbiome | From enrollment to 6 months of age
  The composition of breast milk's microbiome when the child is 2 and 6 months of age
Hormonal levels | From enrollment to 6 months of age
  Child's hormonal levels (testosterone, sex hormone-binding globulin, luteinizing hormone and follicle-stimulating hormone) at birth and at the age of 2 and 6 months
Inflammatory markers | From enrollment to 6 months of age
  Systemic inflammation markers (cytokines, C-reactive protein, soluble urokinase-type plasminogen activator receptor and haptoglobulin) at birth and at the age of 2 and 6 months
Respiratory tract infections | From enrollment to 24 months of age
  Respiratory tract infections by the age of 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Turku University Hospital and University of Turku, Turku, Valitse Maakunta., Finland

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared for research purposes upon special request to the PI
Supporting Information: Study Protocol